CLINICAL TRIAL: NCT02439164
Title: Cohort Study of Sedatives' Effects on Neurological Function in Patients With Eloquent Area Glioma: Comparison With a Control Group Without Intracranial Pathology
Brief Title: Sedatives' Effects on Neurological Function in Patients With Eloquent Area Glioma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Nan Lin, M.D., Beijing Tiantan Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2014MP06
Record Dates: First submitted 2015-04-22; First posted 2015-05-08 (Estimated); Results first posted 2017-08-25 (Actual); Last update posted 2017-08-25 (Actual); Status verified 2017-07

CONDITIONS: Glioma
Keywords: sedation; eloquent area glioma; neurologic function
MeSH Terms: conditions — Glioma | interventions — Midazolam

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Glioma group (Experimental): Patients in this group will be administered sedatives (midazolam or propofol or dexmedetomidine) titrating to mild sedation.
  Interventions: Drug: Midazolam
- non-neurosurgical group (Active Comparator): patients in this group will be administered the same sedative midazolam as compared glioma group, and titrate to mild sedation.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Midazolam — specific benzodiazepine agonist midazolam will be used titrate to desired sedation level, its specific antagonist flumazenil will also be used

SUMMARY:
Sedation in the operating room, the Post Anesthesia Care Unit and the Intensive Care Unit is common and often necessary for patients with intracranial brain tumor. Repeated neurological function assessments is needed in those locations, especially in patients with tumors in or near eloquent regions, this is to monitor their neurologic performance to determine if there are alterations that require treatment. Some slowly infiltrative low-grade gliomas near eloquent regions do not show any detectable neurologic deficits, perhaps from reorganization, but with sedation by some sedatives such as benzodiazepine midazolam and anesthetic hypnotic propofol, the disease may seem much worse resulting in inappropriately aggressive treatment. This may be especially problematic in patients undergoing awake craniotomy for tumors in eloquent regions.

This is a single-center perspective study. Patients will be mildly sedated to keep them responsive and cooperative. Motor and sensory function will be evaluated before and after mild sedation. Specific benzodiazepine antagonist will be used if sedated by midazolam.

The purpose of this study is to observe if commonly used benzodiazepine midazolam exacerbates or unmasks motor and sensory function in patients with intracranial eloquent area gliomas.

Hypothesis:

mild sedation can unmasks or exacerbate motor and sensory deficits in patients with eloquent area glioma but not in non-neurosurgical patients/healthy volunteers. If the neurologic deficits induced by benzodiazepine agonist, then can be reversed by flumazenil.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-60 year-old
* American Society of Anesthesiology(ASA) status I~II
* Elective craniotomy patients with supratentorial eloquent glioma diagnosed by MRI (In control group: volunteers without neuro-diseases)

Exclusion Criteria:

* Unable to comprehend and cooperate with the neurologic examination
* Impaired mental status
* Taking sedative drugs in the past 24 hours
* Taking pain reliever in the past 24 hours
* Drug and/or alcohol abuse
* Pregnant and/o lactating women
* Recurrent brain tumors
* Multiple brain tumors
* Accepting radiotherapy or chemotherapy
* Complicated with intracranial trauma and vascular diseases
* Complicated with grand mal epilepsy ( in midazolam group)
* Complicated with neuromuscular diseases
* Complicated with cutaneous paresthesia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2015-05-26 (Actual); Primary Completion 2017-03-21 (Actual); Study Completion 2017-03-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

RESULTS

PARTICIPANT FLOW:
Groups:
- Glioma Group: Patients in this group will be administered sedatives (midazolam or propofol or dexmedetomidine) titrating to mild sedation.
  Midazolam: specific benzodiazepine agonist midazolam will be used titrate to desired sedation level, its specific antagonist flumazenil will also be used as a reversal
- Non-neurosurgical Group: patients in this group will be administered the same sedative midazolam as compared glioma group, and titrate to mild sedation.
  Midazolam: specific benzodiazepine agonist midazolam will be used titrate to desired sedation level, its specific antagonist flumazenil will also be used as a reversal
Period: Overall Study
Arm/Group | Glioma Group | Non-neurosurgical Group
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: One patient in non-neurosurgical group was dropped out because he reported his carotid disease history after the task testing. In glioma group, pathological diagnosis displayed two with metastasis and one with meningioma, which were excluded during follow-up. There are 15 in the glioma group and 17 in the control group for the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Glioma Group | Non-neurosurgical Group | Total
Number analyzed (Participants) | 15 | 17 | 32
Age, Continuous [Mean (Standard Deviation); unit: years old] | 46 (9) | 35 (7) | 40 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 7 | 7 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 15 | 17 | 32
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 15 | 17 | 32
weight [Mean (Standard Deviation); unit: kg] | 64.9 (14.0) | 75.8 (5.1) | 70.7 (21.1)
education [Count of Participants; unit: Participants]
  primary school | 2 | 3 | 5
  middle school | 2 | 2 | 4
  high school | 8 | 2 | 10
  college | 3 | 10 | 13

OUTCOME MEASURES:

1. Primary Outcome: Task Completing Time Change Between Sedation and Baseline Measured by 9-hole Peg Test
Description: this is a focal neurologic deficits induced by sedatives, the outcome is the performing time changes after sedation as : sedation-baseline.
Time Frame: after sedation
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Glioma Group: Patients in this group will be administered sedative midazolam titrating to mild sedation.
  Midazolam: specific benzodiazepine agonist midazolam will be used titrate to desired sedation level, its specific antagonist flumazenil will also be used as a reversal
Arm/Group | Glioma Group | Non-neurosurgical Group
Number analyzed (Participants) | 15 | 17
seconds
  baseline for contralesional hand | 27.8 (15.9) | 19.1 (3.2)
  after sedation for contralesional hand | 54.3 (32.4) | 21.4 (3.41)
  baseline for ipsilesional hand | 21.8 (7.1) | 19.1 (3.2)
  after sedation for ipsilesional hand | 35.5 (16.6) | 21.4 (3.41)
Statistical Analysis 1: Comparison: Glioma Group vs Non-neurosurgical Group; Test type: Superiority; p < 0.01, t-test, 2 sided; bonferroni correction was used for post hoc analysis, P value less than 0.05 indicated statistical significance; Mean Difference (Net) = 23.51, 95% CI 2-sided [14.16 to 32.87] — this described the difference during midazolam sedation between the glioma and control group without dividing into subgroups; Oneway Analysis of Variance (ANOVA) was used to test the difference among hands in a certain time point. General linear model for repeated measures ANOVA was used to analyze the time difference of test before and after drug administration,

2. Secondary Outcome: Number of Participants With OAA/S=4 After Sedation
Description: OAA/S is Observer Assessment of Sedation with 5 levels (5 = alert, 4 = lethargic, 3 = aroused by voice, 2 = aroused by shaking, 1 = deep sleep), all participants have to achieve OAA/S=4 after sedation.
Time Frame: withing 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Glioma Group | Non-neurosurgical Group
Number analyzed (Participants) | 15 | 17
Participants | 15 | 17

3. Secondary Outcome: Mean Arterial Blood Pressure (MAP) as a Measure of Physiological Change
Description: The MAP was measured at three time points: baseline, sedation and sedation reversal.
Time Frame: 1 hour
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Glioma Group | Non-neurosurgical Group
Number analyzed (Participants) | 15 | 17
mmHg
  baseline MAP | 96.5 (13.5) | 95.7 (14.7)
  sedation MAP | 96.2 (9.5) | 91.2 (12.2)
  sedation reversal MAP | 95.4 (13.6) | 88.2 (14.1)

4. Secondary Outcome: Heart Rate as a Measure of Physiological Change
Description: The HR was measured at three time points: baseline, sedation and sedation reversal.
Time Frame: 1 hour
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Glioma Group | Non-neurosurgical Group
Number analyzed (Participants) | 15 | 17
bpm
  baseline | 78.1 (15.6) | 79.0 (9.1)
  sedation | 84.3 (14.3) | 79.0 (9.4)
  sedation reversal | 81.5 (17.7) | 71.5 (8.9)

5. Secondary Outcome: Brain Glioma Pathological Diagnose as a Measure of Tumor Type
Description: the WHO grade and the type of glioma (WHO glioma grade I~II is regarded as low grade glioma, WHO glioma grade III~IV is regarded as high grade glioma)
Time Frame: 2 weeks
Population: In non-neurosurgical group, patients were not diagnosed as glioma, so the belowed "outcome measure data table" could not indicate the number of glioma grade.
Measure: Count of Participants; unit: Participants
Arm/Group | Glioma Group
Number analyzed (Participants) | 15
Participants
  low grade glioma | 6
  high grade glioma | 9

ADVERSE EVENTS:
Time Frame: 1 hour
Arm/Group | Glioma Group | Non-neurosurgical Group
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/17
Other Adverse Events (participants affected / at risk) | 0/15 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-04-01): https://cdn.clinicaltrials.gov/large-docs/64/NCT02439164/Prot_000.pdf
  • Statistical Analysis Plan (2016-04-01): https://cdn.clinicaltrials.gov/large-docs/64/NCT02439164/SAP_001.pdf